CLINICAL TRIAL: NCT00459498
Title: Significant Intracellular NIS Protein Associated With Low Levels of NIS Messenger RNA in Malignant Thyroid Tumors
Brief Title: Expression of NIS Protein and mRNA in Thyroid Tumors
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Other Study IDs: PRN736/02
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2007-04

CONDITIONS: Tumors
Keywords: NIS; thyroid adenoma; thyroid cancer; Iodine uptake; expression
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The uptake of iodide by thyroid cells requires the expression of sodium iodide symporter (NIS). Thyroid benign and malignant tumors have low iodide uptake activity. Previous studies of NIS expression with RT-PCR and immunohistochemistry showed divergent data. NIS protein was overexpressed in thyroid cancer. The aim of this study was to investigate the NIS transcript levels and its presence and localization in 30 samples of thyroid tumors (14 benign and 16 malignant) and in their surrounding non-tumoral tissues (NT), by real time RT-PCR and immunohistochemistry, respectively. Our results revealed lower gene expression in 78.6% of the benign tumors and 100% of the carcinomas when compared with the NT samples, using GHPDH as a housekeeping gene. Immunohistochemical staining revealed presence of NIS protein in 100% of the non-tumoral samples, 100% of the benign tumors and 93.75% of the malignant tumors. NIS protein was identified at basolateral membrane in 23.3% of non-tumoral samples, 14.3% of benign and 12.5% of malignant tumors. Stronger cytoplasmatic immunostaining of NIS protein was detected in 64.3% of benign tumors and in 87.5% of malignant tumors when compared to NT. Association between low gene expression and strong cytoplasmatic immunostaining was found in 50% of benign tumors and 87.5% of malignant tumors. We concluded that the reduced NIS gene expression in thyroid tumors associated with strong intracytoplasmatic staining may be due to its incapacity to migrate to cellular membrane.

DETAILED DESCRIPTION:
The aim of this study was to quantify NIS transcript levels by real time PCR and to determine the presence and cellular localization of NIS protein by immunohistochemistry, in benign and malignant thyroid tumor cells and to compare with their paired surrounding non-tumoral cell. NIS expression was also compared to that of the TSHR

ELIGIBILITY:
Inclusion Criteria:

* PAtients with thyroid tumors undergoing surgery for total or partial thyroidectomy

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-04; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana K Sodré, Principal Investigator — University of Sao Paulo; Rosalinda Y Camargo, Study Director — University of Sao Paulo

REFERENCES:
- [Background] Saito T, Endo T, Kawaguchi A, Ikeda M, Katoh R, Kawaoi A, Muramatsu A, Onaya T. Increased expression of the sodium/iodide symporter in papillary thyroid carcinomas. J Clin Invest. 1998 Apr 1;101(7):1296-300. doi: 10.1172/JCI1259. PMID 9525971